CLINICAL TRIAL: NCT00996463
Title: Phase II Open Randomized Clinical & Health Economic Trial Comparing Intralesional Antimony Therapy Versus Wound Care Management in Old World Cutaneous Leishmaniasis Patients in Northern Afghanistan
Brief Title: Rationales for Wound Care Management in Old World Cutaneous Leishmaniasis Patients
Acronym: LEICO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Waisenmedizin e. V. Promoting Access to Essential Medicine (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Heidelberg University (Other); University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Prof. Dr. med. Dr. rer. nat. Kurt-Wilhelm Stahl, Waisenmedizin e.V. - PACEM
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFG 08/002
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2009-10

CONDITIONS: Wound Healing
MeSH Terms: interventions — Antimony Sodium Gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IL SSG (Active Comparator): Intralesional sodium stibogluconate
  Interventions: Drug: Sodium Stibogluconate
- ETC+MWT (Experimental): Electro-thermo-coagulation with subsequent moist wound treatment with DAC N-055 (German officinal drug of the German drug codex)
  Interventions: Procedure: Electro-thermo-coagulation; Drug: DAC N-055
- MWT (Experimental): Moist wound treatment with DAC N-055 (German officinal drug of the German drug codex)
  Interventions: Drug: DAC N-055

INTERVENTIONS:
Procedure: Electro-thermo-coagulation — Electro-thermo-coagulation
  Arms: ETC+MWT
Drug: Sodium Stibogluconate — Intralesional injection of sodium stibogluconate
  Arms: IL SSG
Drug: DAC N-055 — Moist wound treatment with DAC N-055 (German officinal drug of the German drug codex)
  Arms: ETC+MWT; MWT

SUMMARY:
The rationales of a clinical trial comparing intralesional antimonial therapy versus wound care management in patients with old world cutaneous leishmaniasis (OWCL) are the following:

1. The effectiveness of the current mainstay treatment with intralesional antimonials for CL is subject to discussion, especially in L. major lesions which are predominant in Northern Afghanistan
2. The importance of wound care management in patients with OWCL has been emphasized by Gonzalez et al. (2008) and its efficacy is confirmed in the Kabul trial with L. tropica patients.

Parallel to the clinical efficacy the trial investigates the cost-effectiveness and -utility of the treatment options under study.

ELIGIBILITY:
Inclusion Criteria:

1. Present a suspected Old World Cutaneous Leishmaniasis lesion confirmed by Giemsa stained wound smears with no other skin diseases or infections and who
2. Have never been previously treated with antimonial injections or any other form of anti-leishmanial medication.

Exclusion Criteria:

1. Patients with more than one lesion are excluded.
2. Patients with a lesion age of > 3 months are also excluded. The experience of the Kabul trial shows that patients presenting themselves for the first time with a lesion, which is older than three months, have either been pre-treated somewhere else and/or show a poor compliance during the trial.
3. Patients below 12 years of age have to be excluded from the trial, because they cannot fill in the EQ-5D and Skindex questionnaire part of the health economic evaluation.
4. Intralesional antimony injections are too painful for lesions located on the nose, lips or eyes. Therefore, patients presenting these lesions are excluded from the trial.
5. For compliance reasons addicted patients and patients not available for follow-up are exclude from the trial.
6. Patients with major uncontrolled diseases as tuberculosis, diabetes or HIV are excluded from the trial, since their management requires additional co-medications, which may affect wound healing.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Wound closure time | 75 days

SECONDARY OUTCOMES:
Leishmania load parasites per gram of tissue before and after treatment | 75 days
Cost-effectiveness & -utility | 75 days

CONTACTS AND LOCATIONS:
Locations (1):
- Leishmaniasis and Malaria Center, Mazari Sharif, Balkh, Afghanistan

REFERENCES:
- [Derived] Stahl HC, Ahmadi F, Schleicher U, Sauerborn R, Bermejo JL, Amirih ML, Sakhayee I, Bogdan C, Stahl KW. A randomized controlled phase IIb wound healing trial of cutaneous leishmaniasis ulcers with 0.045% pharmaceutical chlorite (DAC N-055) with and without bipolar high frequency electro-cauterization versus intralesional antimony in Afghanistan. BMC Infect Dis. 2014 Nov 25;14:619. doi: 10.1186/s12879-014-0619-8. PMID 25420793